CLINICAL TRIAL: NCT04859790
Title: Acceptability/Feasibility Testing of a Virtual Intervention Targeting Anxiety Sensitivity Social Concern
Brief Title: Acceptability/Feasibility Testing of SCAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ohio University (Other)
Responsible Party: Principal Investigator, Nicholas Allan, Assistant Professor of Clinical Psychology, Ohio University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OWG_SCAR INTERVENTION
Record Dates: First submitted 2021-04-01; First posted 2021-04-26 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Social Anxiety

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to the active condition or a waitlist control condition. Participants assigned to the active condition will complete baseline measures and receive the SCAR intervention. They would then complete follow-up measures one month after they completed the SCAR intervention.
  Participants assigned to the waitlist control condition will complete baseline measures and follow-up measures after a month. They will be offered the SCAR intervention after they complete the follow-up measures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active SCAR Intervention (Active Comparator): In this arm, participants will complete baseline measures, receive the SCAR intervention, and complete follow-up measures one month following the intervention.
  Interventions: Behavioral: Social Concerns Appraisal Retraining
- Waitlist Control (No Intervention): Participants assigned to the waitlist control condition will complete baseline measures and measures one month following their baseline appointment. After they complete the follow-up measures, they will be offered the SCAR intervention.

INTERVENTIONS:
Behavioral: Social Concerns Appraisal Retraining — SCAR consists of an hour-long intervention session, followed by a 2-week-long EMI. During the hour-long intervention session, participants will receive psychoeducation (e.g., defining common terms like anxiety), discuss popular misconceptions they may have about publicly observable anxiety symptoms (e.g., "people can tell I'm anxious by looking at me"), and complete exposure exercises (e.g., practicing facing feared physical sensations such as sweating). During the EMI, participants will report on their social anxiety symptoms four times per day. When participants endorse elevated social anxiety during this time, they will receive a targeted message reminding them of the topics covered in the intervention session.
  Arms: Active SCAR Intervention

SUMMARY:
Social anxiety disorder (SAD) is a prominent mental health burden, affecting more than 24 million Americans annually. Social anxiety is worsened by social isolation and severe, ongoing stress. Therefore, it is expected that the COVID-19 pandemic will significantly increase social anxiety symptoms and related impairment. Left untreated, social anxiety typically has a chronic course and a substantial impact on wellbeing. Despite the considerable impact of social anxiety, treatment for social anxiety is underutilized compared to other anxiety disorders, likely due to the distress socially anxious individuals experience upon presenting to treatment. Thus, treatments that are accessible and effective in treating social anxiety are needed. One potential to augment existing treatments for SAD is to develop brief, single-session interventions that could be administered virtually. These interventions could then be combined with additional technological innovations, such as ecological momentary intervention (EMI), to reduce social anxiety. Further, interventions targeting causal risk factors for social anxiety may be particularly beneficial, as these approaches could be used in both prevention and treatment efforts. One risk factor that represents an ideal target for interventions is anxiety sensitivity social concerns (ASSC), defined as the fear of publicly observable symptoms of anxiety (i.e., blushing, trembling, sweating). Although ASSC has been shown to be a risk factor for social anxiety, no interventions have been developed to target ASSC. In the proposed study, a brief (1 hour) virtual intervention targeting ASSC using Cognitive-Behavioral Therapy (CBT) techniques will be developed through examining the acceptability and feasibility of the SCAR intervention prototype. The proposed project holds the promise of developing an intervention to reliably reduce the impact of ASSC, both as a standalone intervention and in combination with other therapeutic approaches.

DETAILED DESCRIPTION:
Social anxiety disorder (SAD) is a mental health disorder characterized by maladaptive distress, anxiety, and avoidance in social situations. Approximately 11% of the United States population will develop SAD in their lifetime, making SAD one of the most prevalent anxiety disorders. SAD is associated with impairment in occupational, social, and familial domains, representing a substantial economic and public health burden. Social anxiety is exacerbated by social isolation , so the effect of social anxiety has likely worsened following the COVID-19 pandemic. Despite the impact of SAD, fewer individuals seek treatment for social anxiety when compared to other common forms of mental illness (e.g., depression) even though effective treatments for social anxiety exist. To increase treatment utilization, brief interventions that target social anxiety-relevant constructs must be developed, as these interventions may be seen as more palatable among socially anxious individuals than the traditional course of treatment for SAD (lasting between 8-12 weekly 1-hour sessions). Additionally, such interventions can be easily administered virtually, reducing risk of COVID-19 transmission.

Causal risk factors, defined as risk factors where a manipulation of the risk factor produces changes in the outcome, represent ideal targets for intervention. To be causal, a risk factor must concurrently relate to and longitudinally predict changes in the outcome. In addition, this risk factor must be malleable; that is, that it can change over time. Developing interventions targeting causal risk factors is an important area of research, as such interventions can both help prevent the development of mental illness and treat mental illness once it has developed. However, limited interventions have been developed that specifically target causal risk factors for social anxiety.

One causal risk factor that may represent an ideal target for interventions is anxiety sensitivity social concerns (ASSC), defined as the fear of publicly observable symptoms of anxiety (e.g., blushing, trembling, sweating). ASSC is one of three dimensions of anxiety sensitivity (AS), which is the overall fear of physiological symptoms of anxiety. The other two dimensions of AS are AS physical concerns (ASPC), defined as the fear of symptoms of anxious arousal (e.g., elevated heart rate, difficulty breathing), and AS cognitive concerns (ASCC), defined as the fear of cognitive dyscontrol (e.g., racing thoughts, feeling "spacy"). The AS dimensions relate thematically to mental illness, with ASSC relating to social anxiety, ASPC relating to panic disorder, and ASCC relating to depression. There are brief interventions targeting overall AS and ASCC; however, no intervention targeting ASSC has been established. Given the link between ASSC and social anxiety, a brief intervention targeting ASSC will likely result in subsequent reductions in social anxiety.

Objectives - Consistent with recommendations for the iterative process of intervention development the current study is designed to 1) gain shareholder feedback to refine an ASSC intervention prototype, termed the Social Concerns Appraisal Retraining (SCAR) and 2) examine acceptability and feasibility ratings for SCAR. The treatment effects of the SCAR intervention on social anxiety will also be examined. However, this will be an exploratory objective, as it is recommended to first develop acceptable and feasible interventions prior to conducting clinical trials to examine treatment effects. The final version of SCAR will consist of an hour-long intervention component, followed by a two-week-long ecological momentary intervention (EMI) component (detailed below). SCAR will be offered to clients of the Ohio University Psychology and Social Work Clinic. Grant funds will be used to cover clinic costs so that SCAR will be made available to 36 clients at the Ohio University Psychology and Social Work Clinic free of charge.

Materials and Methods - The SCAR intervention was developed by adapting previous cognitive-behavioral therapy (CBT)-based AS interventions. In line with previous AS interventions, SCAR will consist of providing psychoeducation (e.g., defining common terms like anxiety), myth busting popular misconceptions clients may have about publicly observable anxiety symptoms (e.g., "people can tell I'm anxious by looking at me"), and completing exposure exercises (e.g., practicing facing feared physical sensations such as sweating). The SCAR intervention will be made available to clients at the Ohio University Psychology and Social Work Clinic as a pilot clinical trial. Interested clients will be randomly assigned to receive SCAR or be placed on a waitlist (for control). For participants assigned to SCAR, directly following the hour-long intervention session, they will complete a 2-week long EMI component in which they report on their social anxiety symptoms four times per day. When participants endorse elevated social anxiety during this time, they will receive a targeted message reminding them of the topics covered in SCAR. Ratings of ASSC and social anxiety will be assessed prior to receiving SCAR, after the intervention session, at the end of the EMI component, and 1-month post intervention. These ratings will be compared to those obtained in the waitlist control group. Participants assigned to the waitlist control group will complete baseline measures and measures a month after their baseline appointment. After participants in the waitlist control group complete the 1-month measures, they will be offered SCAR free of charge.

Significance - The proposed study is designed to develop the first brief intervention targeting ASSC. ASSC is a causal risk factor for SAD, a chronic mental health condition that has a substantial impact on public health. Once developed, SCAR will be used in conjunction with treatments for SAD and in prevention efforts among individuals at risk for developing SAD.

ELIGIBILITY:
Inclusion Criteria:

* Score ≥ 6 on the social concerns subscale of the Anxiety Sensitivity Index-3 OR score ≥ 2 on the Social Phobia Scale-6

Exclusion Criteria:

* Suicidal ideation indicative of a need for hospitalization
* Uncontrolled manic or psychotic-spectrum symptoms
* Not having internet access or owning a smartphone
* Not fluent English speaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Client Satisfaction Questionnaire-8 | Directly following the intervention
  An average Client Satisfaction Questionnaire-8 rating of > 3 (on a 4-point scale) for a study component will provide support for the acceptability and feasibility of this intervention. Scores range from 8-32 with higher scores indicating greater satisfaction.
Client Satisfaction Questionnaire-8 | One month post intervention.
  An average Client Satisfaction Questionnaire-8 rating of > 3 (on a 4-point scale) for a study component will provide support for the acceptability and feasibility of this intervention. Scores range from 8-32 with higher scores indicating greater satisfaction.
Ecological Momentary Intervention Completion Rate | The Ecological Momentary Intervention will directly follow the intervention. Prompts will be delivered four times per day for two weeks.
  The percentage of completed ecological momentary intervention prompts will be used as a measure of acceptability and feasibility. The Ecological Momentary Intervention will be considered feasible if > 80 percent of the Ecological Momentary Intervention sessions are completed by > 80 percent of participants, as done in previous studies (LaFreniere & Newman, 2016; Lucas-Thompson et al., 2019).

SECONDARY OUTCOMES:
Anxiety Sensitivity Index-3 | Before the intervention
  Anxiety Sensitivity Index-3 - 18-item measure assessing anxiety sensitivity. Scores range from 0-72 with higher scores indicating more anxiety sensitivity
Anxiety Sensitivity Index-3 | Directly following the intervention
  Anxiety Sensitivity Index-3 - 18-item measure assessing anxiety sensitivity. Scores range from 0-72 with higher scores indicating more anxiety sensitivity
Anxiety Sensitivity Index-3 | One month post intervention
  Anxiety Sensitivity Index-3 - 18-item measure assessing anxiety sensitivity. Scores range from 0-72 with higher scores indicating more anxiety sensitivity
Social Phobia Scale-6 | Before the intervention
  Social Phobia Scale-6 - 6-item measure assessing social anxiety. Scores range from 0-24 with higher scores indicating more social anxiety
Social Phobia Scale-6 | Directly following the intervention
  Social Phobia Scale-6 - 6-item measure assessing social anxiety. Scores range from 0-24 with higher scores indicating more social anxiety
Social Phobia Scale-6 | One month post intervention.
  Social Phobia Scale-6 - 6-item measure assessing social anxiety. Scores range from 0-24 with higher scores indicating more social anxiety
Social Interaction Anxiety Scale-6 | Before the intervention
  Social Interaction Anxiety Scale-6 - 6-item measure assessing social anxiety. Scores range from 0-24 with higher scores indicating more social anxiety
Social Interaction Anxiety Scale-6 | Directly following the intervention
  Social Interaction Anxiety Scale-6 - 6-item measure assessing social anxiety. Scores range from 0-24 with higher scores indicating more social anxiety
Social Interaction Anxiety Scale-6 | One month post intervention.
  Social Interaction Anxiety Scale-6 - 6-item measure assessing social anxiety. Scores range from 0-24 with higher scores indicating more social anxiety

OTHER OUTCOMES:
Intolerance of Uncertainty Scale-12 | Before the intervention
  Intolerance of Uncertainty Scale-12 - 12-item measure assessing intolerance of uncertainty. Scores range from 12-60 with higher scores representing more intolerance of uncertainty
Intolerance of Uncertainty Scale-12 | Directly following the intervention
  Intolerance of Uncertainty Scale-12 - 12-item measure assessing intolerance of uncertainty. Scores range from 12-60 with higher scores representing more intolerance of uncertainty
Intolerance of Uncertainty Scale-12 | one month post intervention.
  Intolerance of Uncertainty Scale-12 - 12-item measure assessing intolerance of uncertainty. Scores range from 12-60 with higher scores representing more intolerance of uncertainty
Patient Health Questionnaire-9 | Before the intervention
  Patient Health Questionnaire-9 - 9-item measure assessing depression symptoms. Scores range from 0-27 with higher scores representing more depressive symptoms
Patient Health Questionnaire-9 | directly following the intervention
  Patient Health Questionnaire-9 - 9-item measure assessing depression symptoms. Scores range from 0-27 with higher scores representing more depressive symptoms
Patient Health Questionnaire-9 | one month post intervention.
  Patient Health Questionnaire-9 - 9-item measure assessing depression symptoms. Scores range from 0-27 with higher scores representing more depressive symptoms
Brief Penn State Worry Questionnaire | Before the intervention
  Brief Penn State Worry Questionnaire - 5-item measure assessing worry symptoms. Scores range from 5-25 with higher scores indicating more worry.
Brief Penn State Worry Questionnaire | directly following the intervention
  Brief Penn State Worry Questionnaire - 5-item measure assessing worry symptoms. Scores range from 5-25 with higher scores indicating more worry.
Brief Penn State Worry Questionnaire | one month post intervention.
  Brief Penn State Worry Questionnaire - 5-item measure assessing worry symptoms. Scores range from 5-25 with higher scores indicating more worry.
Attentional Control Scale - Straightforward | Before the intervention
  Attentional Control Scale - Straightforward - 20-item measure assessing attentional control. Scores range from 20-80 with higher scores representing better control over attention.
Attentional Control Scale - Straightforward | directly following the intervention
  Attentional Control Scale - Straightforward - 20-item measure assessing attentional control. Scores range from 20-80 with higher scores representing better control over attention.
Attentional Control Scale - Straightforward | one month post intervention.
  Attentional Control Scale - Straightforward - 20-item measure assessing attentional control. Scores range from 20-80 with higher scores representing better control over attention.
Brief Fear of Negative Evaluation-II | Before the intervention
  Brief Fear of Negative Evaluation-II - 12-item measure assessing fear of negative evaluation. Scores range from 12-60 with higher scores representing more fear of negative evaluation.
Brief Fear of Negative Evaluation-II | directly following the intervention
  Brief Fear of Negative Evaluation-II - 12-item measure assessing fear of negative evaluation. Scores range from 12-60 with higher scores representing more fear of negative evaluation.
Brief Fear of Negative Evaluation-II | one month post intervention.
  Brief Fear of Negative Evaluation-II - 12-item measure assessing fear of negative evaluation. Scores range from 12-60 with higher scores representing more fear of negative evaluation.
Panic Disorder Severity Scale | Before the intervention
  Panic Disorder Severity Scale - 7-item measure assessing panic disorder symptoms. Scores range from 0-28 with higher scores indicating more symptoms of panic disorder.
Panic Disorder Severity Scale | directly following the intervention
  Panic Disorder Severity Scale - 7-item measure assessing panic disorder symptoms. Scores range from 0-28 with higher scores indicating more symptoms of panic disorder.
Panic Disorder Severity Scale | one month post intervention.
  Panic Disorder Severity Scale - 7-item measure assessing panic disorder symptoms. Scores range from 0-28 with higher scores indicating more symptoms of panic disorder.
Alcohol Use Disorders Identification Test | Before the intervention
  Alcohol Use Disorders Identification Test - 10-item measure assessing alcohol use disorder symptoms. Scores range from 0-40 with higher scores indicating more symptoms of alcohol use disorder
Alcohol Use Disorders Identification Test | directly following the intervention
  Alcohol Use Disorders Identification Test - 10-item measure assessing alcohol use disorder symptoms. Scores range from 0-40 with higher scores indicating more symptoms of alcohol use disorder
Alcohol Use Disorders Identification Test | one month post intervention.
  Alcohol Use Disorders Identification Test - 10-item measure assessing alcohol use disorder symptoms. Scores range from 0-40 with higher scores indicating more symptoms of alcohol use disorder
Loneliness Questionnaire | Before the intervention
  Loneliness Questionnaire - 5-item measure assessing loneliness. Scores range from 5-25 with higher scores indicating more loneliness.
Loneliness Questionnaire | directly following the intervention
  Loneliness Questionnaire - 5-item measure assessing loneliness. Scores range from 5-25 with higher scores indicating more loneliness.
Loneliness Questionnaire | one month post intervention.
  Loneliness Questionnaire - 5-item measure assessing loneliness. Scores range from 5-25 with higher scores indicating more loneliness.
COVID Behavior Questionnaire | Before the intervention
  COVID Behavior Questionnaire - 12-item measure assessing COVID-19 behaviors. Scores range from 0-48 with higher scores indicating more behaviors due to COVID-19
COVID Behavior Questionnaire | directly following the intervention
  COVID Behavior Questionnaire - 12-item measure assessing COVID-19 behaviors. Scores range from 0-48 with higher scores indicating more behaviors due to COVID-19
COVID Behavior Questionnaire | one month post intervention.
  COVID Behavior Questionnaire - 12-item measure assessing COVID-19 behaviors. Scores range from 0-48 with higher scores indicating more behaviors due to COVID-19
COVID Worry Questionnaire | Before the intervention
  COVID Worry Questionnaire - 12-item measure assessing COVID-19 worries. Scores range from 0-48 with higher scores indicating more worries due to COVID-19
COVID Worry Questionnaire | directly following the intervention
  COVID Worry Questionnaire - 12-item measure assessing COVID-19 worries. Scores range from 0-48 with higher scores indicating more worries due to COVID-19
COVID Worry Questionnaire | one month post intervention.
  COVID Worry Questionnaire - 12-item measure assessing COVID-19 worries. Scores range from 0-48 with higher scores indicating more worries due to COVID-19
Momentary Anxiety Sensitivity Index-3 Social Concerns Subscale | During the Ecological Momentary Intervention portion of the intervention assessed up to 14 days
  Momentary Anxiety Sensitivity Social Concerns - Participants will complete measures assessing momentary experience of anxiety sensitivity social concerns four times per day. Scores range from 0-24 with higher scores indicating more momentary social concerns.
Momentary Social Phobia Scale-6 | During the Ecological Momentary Intervention portion of the intervention assessed up to 14 days
  Momentary Social Phobia Scale-6 - Participants will complete measures assessing momentary experience of social anxiety four times per day. Scores range from 0-24 with higher scores indicating more momentary social anxiety.
Momentary Anxiety Depression Distress Inventory-27 - Anxious Arousal Subscale | During the Ecological Momentary Intervention portion of the intervention assessed up to 14 days
  Momentary Anxiety Depression Distress Inventory-27 - Anxious Arousal Subscale - Participants will complete measures assessing momentary experience of anxious arousal four times per day. Scores range from 0-36 with higher scores indicating more momentary anxious arousal.
Momentary Brief Penn State Worry Questionnaire | During the Ecological Momentary Intervention portion of the intervention assessed up to 14 days
  Momentary Brief Penn State Worry Questionnaire - Participants will complete measures assessing momentary experience of worry four times per day. Scores range from 5-25 with higher scores indicating more momentary worry.

CONTACTS AND LOCATIONS:
Locations (1):
- Ohio University, Athens, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Allan NP, Saulnier KG, Cooper D, Oglesby ME, Schmidt NB. Niacin biological challenge: A paradigm to evaluate social concerns. J Behav Ther Exp Psychiatry. 2019 Dec;65:101489. doi: 10.1016/j.jbtep.2019.101489. Epub 2019 May 30. PMID 31170623
- [Background] Allan NP, Capron DW, Raines AM, Schmidt NB. Unique relations among anxiety sensitivity factors and anxiety, depression, and suicidal ideation. J Anxiety Disord. 2014 Mar;28(2):266-75. doi: 10.1016/j.janxdis.2013.12.004. Epub 2013 Dec 27. PMID 24534564
- [Background] Allan NP, Cooper D, Oglesby ME, Short NA, Saulnier KG, Schmidt NB. Lower-order anxiety sensitivity and intolerance of uncertainty dimensions operate as specific vulnerabilities for social anxiety and depression within a hierarchical model. J Anxiety Disord. 2018 Jan;53:91-99. doi: 10.1016/j.janxdis.2017.08.002. Epub 2017 Aug 7. PMID 28807519
- [Background] Butler AC, Chapman JE, Forman EM, Beck AT. The empirical status of cognitive-behavioral therapy: a review of meta-analyses. Clin Psychol Rev. 2006 Jan;26(1):17-31. doi: 10.1016/j.cpr.2005.07.003. Epub 2005 Sep 30. PMID 16199119
- [Background] Chow PI, Fua K, Huang Y, Bonelli W, Xiong H, Barnes LE, Teachman BA. Using Mobile Sensing to Test Clinical Models of Depression, Social Anxiety, State Affect, and Social Isolation Among College Students. J Med Internet Res. 2017 Mar 3;19(3):e62. doi: 10.2196/jmir.6820. PMID 28258049
- [Background] Drummond PD, Lazaroo D. The effect of niacin on facial blood flow in people with an elevated fear of negative evaluation. Eur Neuropsychopharmacol. 2012 Mar;22(3):200-4. doi: 10.1016/j.euroneuro.2011.07.013. PMID 21856131
- [Background] Keller MB. The lifelong course of social anxiety disorder: a clinical perspective. Acta Psychiatr Scand Suppl. 2003;(417):85-94. doi: 10.1034/j.1600-0447.108.s417.6.x. PMID 12950439
- [Background] Kelly PJ, Kyngdon F, Ingram I, Deane FP, Baker AL, Osborne BA. The Client Satisfaction Questionnaire-8: Psychometric properties in a cross-sectional survey of people attending residential substance abuse treatment. Drug Alcohol Rev. 2018 Jan;37(1):79-86. doi: 10.1111/dar.12522. Epub 2017 May 7. PMID 28480521
- [Background] Kessler RC, Aguilar-Gaxiola S, Alonso J, Chatterji S, Lee S, Ormel J, Ustun TB, Wang PS. The global burden of mental disorders: an update from the WHO World Mental Health (WMH) surveys. Epidemiol Psichiatr Soc. 2009 Jan-Mar;18(1):23-33. doi: 10.1017/s1121189x00001421. PMID 19378696
- [Background] LaFreniere LS, Newman MG. A BRIEF ECOLOGICAL MOMENTARY INTERVENTION FOR GENERALIZED ANXIETY DISORDER: A RANDOMIZED CONTROLLED TRIAL OF THE WORRY OUTCOME JOURNAL. Depress Anxiety. 2016 Sep;33(9):829-39. doi: 10.1002/da.22507. Epub 2016 Apr 7. PMID 27062682
- [Background] Naragon-Gainey K. Meta-analysis of the relations of anxiety sensitivity to the depressive and anxiety disorders. Psychol Bull. 2010 Jan;136(1):128-50. doi: 10.1037/a0018055. PMID 20063929
- [Background] Onken LS, Carroll KM, Shoham V, Cuthbert BN, Riddle M. Reenvisioning Clinical Science: Unifying the Discipline to Improve the Public Health. Clin Psychol Sci. 2014 Jan 1;2(1):22-34. doi: 10.1177/2167702613497932. PMID 25821658
- [Background] Schmidt NB, Capron DW, Raines AM, Allan NP. Randomized clinical trial evaluating the efficacy of a brief intervention targeting anxiety sensitivity cognitive concerns. J Consult Clin Psychol. 2014 Dec;82(6):1023-33. doi: 10.1037/a0036651. Epub 2014 May 12. PMID 24821096
- [Background] Taylor S, Zvolensky MJ, Cox BJ, Deacon B, Heimberg RG, Ledley DR, Abramowitz JS, Holaway RM, Sandin B, Stewart SH, Coles M, Eng W, Daly ES, Arrindell WA, Bouvard M, Cardenas SJ. Robust dimensions of anxiety sensitivity: development and initial validation of the Anxiety Sensitivity Index-3. Psychol Assess. 2007 Jun;19(2):176-88. doi: 10.1037/1040-3590.19.2.176. PMID 17563199
- [Derived] Saulnier KG, Koscinski B, Flynt S, Accorso C, Allan NP. Brief observable anxiety sensitivity treatment: intervention development and a pilot randomized-controlled acceptability and feasibility trial to evaluate a brief intervention for anxiety sensitivity social concerns. Cogn Behav Ther. 2024 Mar;53(2):190-206. doi: 10.1080/16506073.2023.2288551. Epub 2023 Nov 28. PMID 38014462

DOCUMENTS (1):
  • Statistical Analysis Plan (2021-04-21): https://cdn.clinicaltrials.gov/large-docs/90/NCT04859790/SAP_000.pdf